CLINICAL TRIAL: NCT06143748
Title: Cadonilimab Combined With Induction Chemotherapy and Definitive Radiotherapy for Patients With Locally Advanced Esophageal Squamous Cell Carcinoma: a Phase II, Single-arm Trial (EC-CRT-006)
Brief Title: Combination of Cadonilimab and Chemoradiotherapy in Esophageal Cancer (EC-CRT-006)
Acronym: EC-CRT-006
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mian XI, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-425
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Esophagus Cancer
Keywords: Esophageal squamous cell carcinoma; Radiotherapy; Cadonilimab; Induction chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — TP protocol; Paclitaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study group (Experimental): Patients will receive 2 cycles of 3-weekly schedule of induction chemotherapy, consisting of paclitaxel 135 mg/m2, cisplatin 75 mg/m2, and cadonilimab 10 mg/kg on day 1 prior to CRT. Then all patients will receive standard fractionation radiation therapy scheme: 50.4 Gy in 28 fractions, concurrently with 2 cycles of cadonilimab. After the completion of radiotherapy, patients will then receive 12 additional cycles of cadonilimab.
  Interventions: Drug: Cadonilimab; Drug: Paclitaxel and cisplatin; Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Cadonilimab — Patients received cadonilimab 10 mg/kg every 3 weeks for up to 16 cycles.
  Other Names: AK104
Drug: Paclitaxel and cisplatin — Patients received 2 cycles of induction chemotherapy with paclitaxel/cisplatin (paclitaxel 135 mg/m2 and cisplatin 75 mg/m2) prior to radiotherapy. Then patients will not receive chemotherapy during radiotherapy.
  Other Names: taxol, DDP
Radiation: intensity-modulated radiotherapy — All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is 50.4 Gy in 28 fractions over 5-6 weeks.
  Other Names: IMRT

SUMMARY:
Definitive chemoradiotherapy (CRT) is the standard treatment option for unresectable locally advanced esophageal cancer. However, as high as more than 40% of patients with esophageal cancer experienced locoregional recurrence after definitive CRT. Immune checkpoint inhibitors targeting PD-1/PD-L1 and/or CTLA-4 have shown substantial clinical benefits in advanced esophageal cancer. Recently, the combination of immunotherapy with CRT has emerged as a promising strategy to improve clinical outcomes in esophageal cancer. The aim of this study was to evaluate the efficacy and safety of cadonilimab (a bispecific PD-1/CTLA-4 antibody) combined with induction chemotherapy followed by definitive radiotherapy in patients with locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
A total of 46 patients with unresectable, locally advanced ESCC will be enrolled to receive cadonilimab plus induction chemotherapy followed by definitive radiotherapy and then 12 additional cycles of maintenance therapy with cadonilimab.

Patients will receive 2 cycles of 3-weekly schedule of induction chemotherapy, consisting of paclitaxel 135 mg/m2, cisplatin 75 mg/m2, and cadonilimab 10 mg/kg on day 1 prior to CRT. Then all patients will receive standard fractionation radiation therapy scheme: 50.4 Gy in 28 fractions, concurrently with 2 cycles of cadonilimab. After the completion of radiotherapy, patients will then receive 12 additional cycles of cadonilimab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Locally advanced, and absence of distant metastasis disease, confirmed by endoscopic ultrasound (EUS) and PET-CT scan, stage II-IVA (according to UICC TNM version 8);
3. Not suitable for surgery (either for medical reasons or patient's choice);
4. Age at diagnosis 18 to 75 years;
5. No prior cancer therapy;
6. Estimated life expectancy >6 months;
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. No history of concomitant or previous malignancy;
9. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥4.0×109/L, absolute neutrophil count (ANC) ≥1.5×109/L; b. platelets ≥100×109/L; c. hemoglobin ≥9g/dL; d. serum albumin ≥2.8g/dL; e. total bilirubin ≤1.5×ULN, ALT, AST and/or AKP ≤2.5×ULN; f. serum creatinine ≤1.5×ULN or creatinine clearance rate >60 mL/min;
10. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Patients with distant metastasis disease or esophageal fistula at diagnosis;
3. Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of cadonilimab, and the chemotherapeutic drugs paclitaxel or cisplatin;
4. Patients who have a preexisting or coexisting bleeding disorder;
5. Female patients who are pregnant or lactating;
6. Inability to provide informed consent due to psychological, familial, social and other factors;
7. Presence of CTC grade ≥2 peripheral neuropathy;
8. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer
9. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
10. Patients who cannot tolerate chemoradiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia.
11. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
12. A history of interstitial lung disease or non-infectious pneumonia;
13. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of enrollment until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 36 months.
  Three-year follow-up from the date of enrollment to the date of disease progression or last follow-up

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 36 months.
  Three-year follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Clinical complete response | 3 months after radiotherapy (plus or minus 7 days)
  Tumor response was evaluated 3 months after the completion of treatment based on CT or PET-CT scans, and endoscopy with biopsies.
Duration of response | From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 36 months.
  From the date of first CR/PR to the date of first PD.
Treatment-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0.

OTHER OUTCOMES:
Correlation between immune signature and survival | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between pretreatment immune signature (PD-L1, CD8, CTLA-4, CD56, and CD68) by mIHC and survival outcomes.
Correlation between dynamic change of ctDNA and survival | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between dynamic change of ctDNA during treatment and survival outcomes.
Correlation between genetic biomarkers and survival | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between baseline genetic biomarkers by whole-exome sequencing and RNA-sequencing and immune-related adverse event, clinical response, and survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gao X, Xu N, Li Z, Shen L, Ji K, Zheng Z, Liu D, Lou H, Bai L, Liu T, Li Y, Li Y, Fan Q, Feng M, Zhong H, Huang Y, Lou G, Wang J, Lin X, Chen Y, An R, Li C, Zhou Q, Huang X, Guo Z, Wang S, Li G, Fei J, Zhu L, Zhu H, Li X, Li F, Liao S, Min Q, Tang L, Shan F, Gong J, Gao Y, Zhou J, Lu Z, Li X, Li J, Ren H, Liu X, Yang H, Li W, Song W, Wang ZM, Li B, Xia M, Wu X, Ji J. Safety and antitumour activity of cadonilimab, an anti-PD-1/CTLA-4 bispecific antibody, for patients with advanced solid tumours (COMPASSION-03): a multicentre, open-label, phase 1b/2 trial. Lancet Oncol. 2023 Oct;24(10):1134-1146. doi: 10.1016/S1470-2045(23)00411-4. PMID 37797632
- [Result] Frentzas S, Gan HK, Cosman R, Coward J, Tran B, Millward M, Zhou Y, Wang W, Xia D, Wang ZM, Li B, Xia M, Desai J. A phase 1a/1b first-in-human study (COMPASSION-01) evaluating cadonilimab in patients with advanced solid tumors. Cell Rep Med. 2023 Nov 21;4(11):101242. doi: 10.1016/j.xcrm.2023.101242. Epub 2023 Oct 17. PMID 37852261
- [Result] Doki Y, Ajani JA, Kato K, Xu J, Wyrwicz L, Motoyama S, Ogata T, Kawakami H, Hsu CH, Adenis A, El Hajbi F, Di Bartolomeo M, Braghiroli MI, Holtved E, Ostoich SA, Kim HR, Ueno M, Mansoor W, Yang WC, Liu T, Bridgewater J, Makino T, Xynos I, Liu X, Lei M, Kondo K, Patel A, Gricar J, Chau I, Kitagawa Y; CheckMate 648 Trial Investigators. Nivolumab Combination Therapy in Advanced Esophageal Squamous-Cell Carcinoma. N Engl J Med. 2022 Feb 3;386(5):449-462. doi: 10.1056/NEJMoa2111380. PMID 35108470
- [Result] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609